CLINICAL TRIAL: NCT00571870
Title: Study on the Effect of GnRH Antagonist on hCG Day on Outcomes of Controlled Ovarian Hyperstimulation With GnRH Antagonist Flexible Multiple-dose Protocols
Brief Title: Gonadotropin-releasing Hormone Antagonist on Triggering Day: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Chang Suk Suh, Dept. of Obstetrics and Gynecology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-0710-050-001
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Stimulated as conventional protocol
  Interventions: Drug: cetrorelix acetate
- B (Experimental): GnRH antagonist stopped one day earlier than conventional protocol
  Interventions: Drug: cetrorelix acetate

INTERVENTIONS:
Drug: cetrorelix acetate — The GnRH antagonist, cetrorelix acetate (Cetrotide; Serono) 0.25 mg was added daily, starting when the leading follicle reached 14 mm in diameter during ovarian stimulation for IVF. When the leading follicle reached a mean diameter of 18 mm or two follicles or more reached a diameter of 17 mm, 250 μg of recombinant hCG (Ovidrel; Serono) SQ was injected. In Group A, the GnRH antagonist continued to be used until the day of hCG administration. In Group B, the GnRH antagonist was not administrated on the hCG day

SUMMARY:
Gonadotropin-releasing hormone (GnRH) antagonists have been widely used for the prevention of premature luteinizing hormone (LH) surges during controlled ovarian hyperstimulation (COH) for in vitro fertilization and embryo transfer (IVF-ET) since the late 1990's.

Many years have passed since GnRH antagonists were introduced to prevent premature LH surges during stimulated cycles. However, there is still no consensus on the optimal GnRH antagonist protocol. Attempts at modifying GnRH antagonist protocols have been made to improve COH outcomes. However, a meta-analysis of 27 randomized controlled trials, including recent reports, showed significantly lower clinical ongoing pregnancy rates in the antagonist group. Thus, additional efforts are needed to identify the optimal stimulation protocols to achieve better follicular and embryonic development and to improve the pregnancy rates in COH using GnRH antagonist.

Given the assumption of a detrimental effect of GnRH antagonist on the pregnancy rate, with current protocols, we hypothesized that a shorter duration of GnRH antagonist administration might improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Both ovaries present with no morphological abnormalities
* Normal ovulatory cycle with cycle lengths of between 25 and 35 days
* Basal serum FSH (day 3) level of < 15 mIU/mL
* Body mass index (BMI) ranging between 18 and 27 kg/m2

Exclusion Criteria:

* History of a poor ovarian response
* Evidence of endocrine abnormalities, such as, hyperprolactinemia, thyroid dysfunction, or polycystic ovary syndrome
* Hydrosalpinx
* Severe endometriosis (stage III-IV)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maturity of oocytes, fertilization rate, embryo quality | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Chang Suk Suh, M.D., Ph.D., Principal Investigator — Dept. of Obstetrics and Gynecology, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea